CLINICAL TRIAL: NCT02664402
Title: Analysis of A Tool to Assess Psycho Social Spiritual Healing: Cognitive Interviewing
Brief Title: Tool to Assess Psycho-Social-Spiritual Healing: Cognitive Interviewing
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 160056; 16-CC-0056
Record Dates: First submitted 2016-01-26; First posted 2016-01-27 (Estimated); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Palliative Care; Critical Illness
Keywords: Palliative Care; Pain; Community Health; Natural History
MeSH Terms: conditions — Critical Illness; Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults: English speaking, physician diagnosed with a life threatening illness.

SUMMARY:
Background:

People undergo many changes when they have a life-threatening illness. Their values may change. They may have less fear of illness and death. They may become more spiritual. Researchers made a questionnaire called HEALS (Healing Experience During All Life Stressors). They want to use it to better understand these positive changes. They hope to provide better care for people with serious illnesses.

Objectives:

To develop the HEALS tool to better understand psycho-social-spiritual healing in people with serious illnesses. Also, to find out how palliative care services help people handle their illness or stress.

Eligibility:

Adults at least 18 years old at least 91 days after being diagnosed with a life-threatening illness. They must be getting:

Inpatient or outpatient palliative care at NIH Clinical Center OR

Inpatient palliative care at Suburban Hospital OR

NIH outpatient palliative care provided at Mobile Medical Care Clinic

Design:

Participants will be screened with questions to make sure they are eligible.

Participants will have 1 individual research session. This will be at the NIH Clinical Center.

Participants will be interviewed by a research team member. They will be asked about changes in a person s way of living that might happen during or after a serious illness.

Participants will be asked for their thoughts and opinions about the questions. They will be asked what ideas they may have to make the questions better.

Interviews will be audiotaped.

Participants will be asked some questions specific to their care location and team. These are to better understand how their services are helping participants.

...

DETAILED DESCRIPTION:
Background:

We identify healing in the context of chronic or life-threatening illness as a patient-reported outcome consisting of growth or benefit in psychological, social and/or spiritual dimensions representing improvement well above the patient s pre-morbidity baseline. This positive outcome often occurs despite substantial suffering during the illness, even in terminal cases. Current literature reflects numerous studies suggesting that psychological, social, and/or spiritual dimensions influence positive patient health outcomes and affects overall quality of life. This trend parallels a movement to understand how a difficult experience, such as a cancer diagnosis for example, may help facilitate positive growth, also referred to as healing. Although attention to positive growth/healing in the treatment of life limiting illness is increasing, a psychometrically sound instrument that assesses psycho-social-spiritual (PSS) growth as a means to healing does not exist. The ability to assess healing will allow improvements in programs aimed at helping individuals make positive personal changes in their health-related behavior (our larger program on healing). Content analysis of this contributes to construct validity of the assessment and brings us closer to creating a psychometrically sound measure of psycho- social spiritual healing.

This swill use cognitive interviewing to examine item performance of the NIH HEALS Assessment (healing experience during all life stressors) tool.

Objectives:

Primary Objective

* To continue with instrument development of a tool to assess an individual s progression toward psycho-social spiritual healing by evaluating the participant s understanding of questionnaire items through a cognitive interviewing technique.
* Examine differences in the understanding of questionnaire items between the three recruitment sites.

Eligibility:

* Age greater than or equal to 18 years old
* Understand and speak English
* Physician diagnosed with a life threatening illness
* 91+ days post diagnosis of life threatening illness
* Receiving inpatient or/ outpatient palliative care at NIH Clinical Center inpatient palliative Care at Suburban Hospital, and NIH outpatient palliative care provided at the Mobile Medical Care Clinic

Design:

* Exploratory descriptive study using mix-methods
* Cognitive interviews using retrospective probing in a purposive sample with three rounds of 10 for a total maximum sample of 30 participants, with the completion of content analysis after each round of 10 to inform content and clarity of question items.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Adults age greater than or equal to 18 years. The instrument under study for validation in this protocol is a self-assessment specifically designed for adult populations. Adults above the age of 18 are able to use logic, deductive reasoning, think more about the world / environment and has an understanding and ability to apply abstract ideas, which are all necessary for retrospective cognitive processes
* Understand and speak English
* Oriented to person, time and place at time of interview
* Physician diagnosed with life threatening illness
* 91+ days post diagnosis of life threatening illness
* Receiving inpatient or outpatient palliative care at NIH Clinical Center, inpatient palliative Care at Suburban Hospital, and NIH outpatient palliative care provided at the Mobile Medical Care Clinic

EXCLUSION CRITERIA:

* Patients with known brain metastases will be excluded because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of the assessment questions
* Inability to provide informed consent
* Inability to meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A purposive sample of 30 participants were recruited from patients with scheduled appointments at the palliative care clinic or inpatients at 3 locations: l)Mobile Medical Care, Rockville, MD, 2) Suburban Hospital, Bethesda, MD, 3)NIH Clinical Center, Bethesda, MD.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-01-05 (Actual); Primary Completion 2017-01-05 (Actual); Study Completion 2017-01-05 (Actual)

PRIMARY OUTCOMES:
NIH HEALS Assessment | Present
  Newly developed 49-item questionnaire being evaluated for participant understanding of each item included in questionnaire.

SECONDARY OUTCOMES:
Risk Assessment for Barriers to Palliative Care | present
  Questions from this assessment will help healthcare providers complete a needs assessment with the patient and caregiver in order to better understand patient needs and to identify barriers to using palliative care in a low-income population

CONTACTS AND LOCATIONS:
Overall Officials: Ann M Cohen Berger, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Egnew TR. The meaning of healing: transcending suffering. Ann Fam Med. 2005 May-Jun;3(3):255-62. doi: 10.1370/afm.313. PMID 15928230
- [Background] Denz-Penhey H, Murdoch C. Personal resiliency: serious diagnosis and prognosis with unexpected quality outcomes. Qual Health Res. 2008 Mar;18(3):391-404. doi: 10.1177/1049732307313431. PMID 18235162
- [Background] Lyckholm LJ, Coyne PJ, Kreutzer KO, Ramakrishnan V, Smith TJ. Barriers to effective palliative care for low-income patients in late stages of cancer: report of a study and strategies for defining and conquering the barriers. Nurs Clin North Am. 2010 Sep;45(3):399-409. doi: 10.1016/j.cnur.2010.03.007. Epub 2010 May 10. PMID 20804885
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-CC-0056.html